CLINICAL TRIAL: NCT00873717
Title: Improvement of Nutritional Status in Elderly Residents of Long-term Facilities: Impact of Two Strategies (Oral Care and Dietary Control)
Brief Title: Improvement of Nutritional Status in Elderly Residents of Long-term Facilities
Acronym: Nutrident
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AOM07055; K070103 (Other: APHP); 2008-A00039-46 (Other: IDRCB)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2009-04

CONDITIONS: Nutrition Disorders
Keywords: elderly; long-term facilities; nutritional status
MeSH Terms: conditions — Nutrition Disorders | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dentary (Experimental): Intervention: trimestrial follow-up of patients and counseling for appropriate care (if needed), in order to restore a minimum masticatory function, associated with particular focus on the realization of daily oral wash.
  Interventions: Other: Dentary
- Nutrition (Experimental): control of the administration of dietary prescriptions, incitement to eat.
  Interventions: Other: Nutrition
- Dentary + nutrition (Experimental): cleaning-up of oral cavity, with trimestrial dental and oral check-up with counseling for appropriate care (if needed) associated with control of the administration of dietary prescriptions, incitement to eat.
  Interventions: Other: Dentary + Nutrition
- Control (No Intervention): usual care

INTERVENTIONS:
Other: Dentary — cleaning-up of oral cavity, with trimestrial dental and oral check-up with counseling for appropriate care (if needed).
  Arms: Dentary
Other: Nutrition — control of the administration of dietary prescriptions, incitement to eat.
  Arms: Nutrition
Other: Dentary + Nutrition — trimestrial follow-up of patients and counseling for appropriate care (if needed), in order to restore a minimum masticatory function, associated with particular focus on the realization of daily oral wash.
  associated with control of the administration of dietary prescriptions, incitement to eat.
  Other Names: Dentary and Nutrition
  Arms: Dentary + nutrition

SUMMARY:
Elderly persons in long-term facilities often have denutrition, associated with a bad oral and dental status. Yet, many elderly persons don't attend dentist care and when they have dental prothesis, do not often use them during meals. The impact of a rehabilitation of dental function on their nutritional status has not been proven.

The objective of this study is to assess the impact of 2 strategies aimed to restore a good nutritional status, among patients with slight denutrition.

DETAILED DESCRIPTION:
Two interventions are evaluated during a 1 year study period, with a 4 arms factorial design.

The "Dentary" intervention implies a trimestrial follow-up of patients and counseling for appropriate care (if needed), in order to restore a minimum masticatory function, associated with particular focus on the realization of daily oral wash.

The "Nutrition" intervention consists in 1) comparing the meals and oral supplements administered with the dietary prescriptions and 2) Incite patients to eat.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric Nutritional Risk Index = 83.5 to 97.5; minimum age of 70 years old; living in long-term facilities; more than 6 months of anticipated length of stay

Exclusion Criteria:

* refusal to participate in the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
comparison of GNRI mean-score between arms | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CHARRU, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Marysette FOLLIGUET, DDS, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (6):
- France (6):
  - Centre gérontologie Les Abondances, Boulogne-Billancourt, Île-de-France Region
  - Institut ROGUET, Clichy, Île-de-France Region
  - AP-HP, Louis Mourier Hospital, Colombes, Île-de-France Region
  - Hôpital Bretonneau, Paris, Île-de-France Region
  - Hôpital de Puteaux, Puteaux, Île-de-France Region
  - AP-HP, Hôpital René Muret-Bigottini, Sevran, Île-de-France Region